CLINICAL TRIAL: NCT05792683
Title: Comparison of Duration of CSF Leak in Post Traumatic Patients Managed by Early Lumbar Drain vs Conservative Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Dr Atiq ur Rehman, dr atiq, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEHRIA
Record Dates: First submitted 2023-03-01; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: CSF Leakage
MeSH Terms: conditions — Cerebrospinal Fluid Rhinorrhea

STUDY DESIGN:
Intervention Model Description: ramdomized control trail
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early lumbar drain (Active Comparator): 30 in this group
  Interventions: Device: lumbar drain
- conservative treatment (Other): 30 in this group
  Interventions: Device: lumbar drain

INTERVENTIONS:
Device: lumbar drain — Patient will be placed in the lateral decubitus position; catheter will be inserted by using a Tuohy needle in the interspinous area of lumbar spine. The LD catheter will reach the lumbar subarachnoid space.The remaining part of the drainage kit will be placed along the back of the patient. The catheter insertion site will be sutured and treated with povidone-iodine ointment. Sterile drape will be used to cover the entire external part of the LD.
  The CSF will be collected within the closed beg. CSF drainage through LD will be around 10 ml per hour or 200-250 ml/day.

SUMMARY:
As limited data is available locally and internationally regarding early Lumbar drain and its effect on duration of CSF leak we have decided to compare it conservative treatment. By providing CSF an alternative route for drainage, the fistula site will remain dry. Leakage site won't be facing CSF pressure, and this will promote early healing of the wound.

DETAILED DESCRIPTION:
Cerebrospinal fluid (CSF)leak is caused by communication between the subarachnoid space and the air-filled spaces of the middle ear or para nasal sinuses and sometimes skin. CSF leaks can be divided into two types ,traumatic and non traumatic. The traumatic CSF leaks further divided into accidental and iatrogenic (post surgical procedures) 1. Almost 80% of CSF leaks are due to road traffic accidents, fall from heights and firearms injuries to brain and spine, 16% are iatrogenic, and 4% are non-traumatic 1,2. More than 50% of traumatic CSF leaks are evident within the first 02 days, 70% within the first week, and almost all present within the first 3 months [2,3]. It is estimated that in patients with skull base fracture 10-30% develops CSF leaks and 2% of all traumatic head injuries are associated with CSF leaks [4].With the help of conservative treatment most of the CSF leaks stop within 7-10 days 1,5. When the CSF leak doesn't stop after 7-10 days, a lumbar drainage (LD) is suggested3,7. LD(lumbar drain) is a recommended treatment method for the CSF leaks in skull base and spinal trauma, the indications for LD(lumbar drain ) placement are still controversial ,LD(lumbar drain) effect on early CSF leakage cessation is still arguable 2,3. Traumatic CSF leaks duration can be reduced by early( lumbar drain) placement . At tertiary level particularly in public hospital, our study will be helpful to document the benefits of early lumbar drain (LD) in traumatic CSF leakage patients and their hospital stay. This will also help to reduce the ambiguity regarding the protocol for early lumbar drain (LD) placement .

ELIGIBILITY:
Inclusion Criteria:

1. Age between 15-60 years in both genders.
2. Patients with craniospinal post traumatic or post operative CSF leakage for more than 24 hours.

Exclusion Criteria:

1. Patients with comorbid like Cardiovascular, Chronic Kidney Disease, Coagulopathies and Pregnancy
2. Previous history of chest or abdominal surgery.
3. Previous history of any lumbosacral surgery.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-21 (Actual); Primary Completion 2023-07-21 (Estimated); Study Completion 2023-08-21 (Estimated)

PRIMARY OUTCOMES:
Length of active CSF leak in post-traumatic patients with Lumbar drain. | 06 months
  Lumbar drain will reduce the CSF pressure on the wound which will lead to early healing of CSF leak sight.it will reduce the duration of CSF leak in post traumatic patients .

SECONDARY OUTCOMES:
incidence of recurrence of CSF leaks, meningitis after treatment | with in 06 months
  After treatment with both methods the incidence of recurrence of CSF leaks and meningitis will be recorded .

CONTACTS AND LOCATIONS:
Overall Officials: Atiq UR [arehman], Principal Investigator — Rawalpindi Medical College
Locations (1):
- RMU, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Results of study